CLINICAL TRIAL: NCT02718703
Title: Project EV Minus Regulatory Clinical Evaluation - System Accuracy, User Performance and System Use Evaluation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: LifeScan (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None
Other Study IDs: 3129822
Record Dates: First submitted 2016-03-01; First posted 2016-03-24 (Estimated); Last update posted 2016-09-14 (Estimated); Status verified 2016-09

CONDITIONS: Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Blood Glucose monitoring System (BGMS) (Experimental): Intervention: Blood Glucose monitoring System (BGMS) Results obtained from the BGMS for UP and SA are compared to a reference instrument (YSI)
  Interventions: Device: Blood Glucose Monitoring System.

INTERVENTIONS:
Device: Blood Glucose Monitoring System. — In vitro diagnostic medical device

SUMMARY:
Clinical Evaluation including System Accuracy, User Performance and System Use Evaluation of a new Blood Glucose Monitoring System.

ELIGIBILITY:
Summary of Inclusion Criteria:

* Able to voluntarily provide written informed consent to participate in the study.
* User Performance Accuracy Testing Only: Self-Monitoring - Subject is currently performing unassisted self-monitoring of blood glucose.

Exclusion Criteria:

* Female subjects who are pregnant or lactating.
* Subjects who, in the opinion of the Investigator, are unsuitable for participation in the study.
* User Performance Accuracy Testing Only -Prior involvement with the investigational BGMS being used in this study.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 34 (Actual)
Dates: Start 2015-02; Primary Completion 2015-03 (Actual); Study Completion 2015-03 (Actual)

PRIMARY OUTCOMES:
User Performance (UP) evaluation - blood glucose level: BGMS vs reference instrument. | Up to 1 hour
  UP evaluation of blood glucose monitoring systems compared to a reference instrument. Samples collected by subject and HCP ( HealthCare Professional)
System Accuracy (SA) evaluation - blood glucose level: BGMS vs reference instrument. | Up to 1 hour
  Accuracy verification of blood glucose monitoring systems compared to a reference instrument. Samples collected by HCP only.
System Use Evaluation - HCP ( HealthCare Professional) questionnaire | Up to 1 hour
  Assessing use of BGMS and supporting material by subject.

CONTACTS AND LOCATIONS:
Overall Officials: Lorna Stewart, Study Director — LifeScan
Locations (1):
- BioKinetic Europe Ltd, Belfast, Antrim, United Kingdom

IPD SHARING:
Plan to Share IPD: No